CLINICAL TRIAL: NCT02674724
Title: The Effect of Resistance Training on Balance in Patients With Parkinson Disease: A Pilot Study
Brief Title: The Effect of Resistance Training in Parkinson Disease: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Department of Neurology
Record Dates: First submitted 2016-01-14; First posted 2016-02-04 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2016-10

CONDITIONS: Parkinson Disease
Keywords: Resistance Training; Postural Balance; Exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gym Group (Experimental): With gym equipments, twice per week for 12 weeks.
  Interventions: Other: Gym Group
- Free Weights Group (Active Comparator): With dumbbells, elastics, twice per week for 12 weeks.
  Interventions: Other: Free Weights Group
- Control Group (Placebo Comparator): The control group will be instructed to perform stretching exercises at home in the same 12-week period, according to an illustrated booklet.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Gym Group — Patients from Gym Group will perform a strengthening program of 45 minutes sessions, twice a week in a 12-week period.
  The initial load is established as 60% of one-repetition maximum strength test (1RM) applied for each exercise at the beginning of program. Patients will be encouraged to perform 3 sets of 8 to 12 repetitions. All subjects will be instructed to rest for 30-60 second intervals between sets.
  Arms: Gym Group
Other: Free Weights Group — Patients from Free Weights Group will perform a strengthening program of 45 minutes sessions, twice a week in a 12-week period. The program aim to recruit the same muscles requested in Gym Group. Investigators will apply six different exercises with patients lying supine,standing in stance, sitting and in four points kneeling. All exercises aim to strengthen abdominal muscles, trunk extensors, gluteus, quadriceps and scapula adductors. Patients will perform 3 sets of 8 to 12 repetitions, the load will be offered with dumbbells, elastics with different resistances and anklets.
  Arms: Free Weights Group
Other: Control Group — All three groups will be instructed to perform stretching exercises of trunk, leg and shoulder muscles, according to an illustrated booklet. Only the Control Group patients will be instructed to perform stretching exercises at home in the same 12-week period.
  Arms: Control Group

SUMMARY:
To investigate if resistance training exercises performed twice a week with or without gym equipment assistance in a 12-week period could improve balance in patients with Parkinson Disease (PD).

Methods: Sixty three patients with idiopathic PD (Hoehn and Yahr stage II - III) and preserved cognitive function will participate in this study. Patients will be randomized among three intervention groups: resistance training with free weights, resistance training with gym equipment and control group. Investigators will use static platform balance variables to assess the primary end-point outcome measures. For the secondary outcomes measures, most common clinical functional balances tests for PD will be applied: Berg Balance Scale (BBS), Mini-BESTest - Balance Evaluation (Mini-BESTest), Timed Up and Go test (TUG) and variables from dynamic posturography.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurodegenerative disease that affects motor functions and is characterized by bradykinesia, resting tremor, rigidity, and postural instability. Despite of pharmacological treatments, patients remain with deficits in balance, gait, autonomic system functions and cognition which impact on their quality of life.

The effects of resistance training on PD are still controversial when balance and improvement on functional tests are the targets.

Since the results of previous studies about resistance training on balance are still controversial, more interventions are required to address the question if strengthening exercise may improve or not the balance of PD patients. Our exercises will target the trunk, leg and shoulder muscles because of their contribution on patient's posture.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 to 75 years old;
* Hoehn and Yahr stages II or III;
* Idiopathic Parkinson disease diagnosed according to the United Kingdom Parkinson's Disease Society Brain Research Centre Criteria, Institute of Neurology, London;
* Ability to walk independently without walking devices aid;
* Absence of orthopedic injuries or pain in joints that could interfere on training program;
* Stable medication regimen for PD treatment at recruitment stage;
* Mini Mental State Examination Scale (MMSE) ≥ to 27 for literate patients and schooling ≥ of 4 years of formal education;
* No cardiovascular instability;
* No pacemaker, decompensated metabolic disease, vestibular dysfunction, and stroke;
* Availability to come to the clinic twice a week;
* Not participating in other physical rehabilitation programs during and six months prior to the study.

Exclusion Criteria:

* Patients will be excluded if they refuse to participate, do not sign the consent form, have a diagnosis of secondary parkinsonism or present cognitive impairment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-05 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Postural sway on Static Posturography | 12 weeks
  Static Posturography is a technique used to objectively assess postural sway with patients standing still on a fixed platform that measures center of pressure displacement. Tests were standardized such as the feet position, the eye gaze and environment light, with three trials of 60-second test in eyes - open, eyes closed and eyes open in dual task condition. Investigators will analyze the anteroposterior displacement, medial-lateral displacement, area, velocity and path length.

SECONDARY OUTCOMES:
Balance on Berg Balance Scale | 12 weeks
  Berg Balance Scale is used to assess balance and falls in elderly using different tasks. It consists of 14 tasks scoring from zero to four, zero means that the patient is unable to perform the task and four means that the task is performed independently.
Balance Evaluation on Mini-BESTest | 12 weeks
  The Mini-BESTest contains 14 items that assess dynamic balance focusing on anticipatory postural adjustments, postural responses, sensory orientation and stability in gait. Items are scored from 0 to 2 (normal performance in balance).
Functional balance and gait on Timed Up and Go test (TUG) | 12 weeks
  The TUG test measures individual speed while performing the sequence: rising from a chair, walking for three meters of distance, turning around and returning to the starting position, sitting on a chair. When the examination exceeds 13 seconds, patients have higher risk of falls.
Quality of life on PDQ-39 Questionnaire | 12 weeks
  The PDQ-39 assess quality of life of Parkinson's disease patients over the last month. Contains 39 items and eight dimensions (Mobility, Activities of daily living, Emotional well-being, Stigma, Social support, Cognitions and Bodily discomfort).
Functional balance on Dynamic Posturography | 12 weeks
  Dynamic posturography is a quantitative method to assess balance. This system have sensors located below two platforms and measures vertical and horizontal forces produced by the center of gravity during a pre-determined task (sit to stand, tandem walk and step over).

CONTACTS AND LOCATIONS:
Overall Officials: Egberto Reis Barbosa, MD, PhD, Study Director — Department of Neurology, Clinics Hospital of University of São Paulo Faculty of Medicine, São Paulo, Brazil.
Locations (1):
- Department of Neurology of University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886